CLINICAL TRIAL: NCT03539237
Title: Effect of an Intensity Level Video Demonstration on the Gap Between Self-reported and Accelerometer-measured Physical Activity in Individuals Aged 40 to 75 Years
Brief Title: Closing the Gap Between Self-reported and Accelerometer-based Physical Activity
Acronym: GAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: GAP05/18
Record Dates: First submitted 2018-05-15; First posted 2018-05-29 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Physical Activity
Keywords: Video demonstration; Intensity levels; Physical activity; Self-report; Accelerometer
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Video"-group (Experimental): Video group: Individuals in this group receive the intervention "Video demonstration of physical activity intensity levels". They watch a 3-minute-video explaining and visualizing light-, moderate-, and vigorous-intensity levels of physical activity before completing a tablet PC-supported physical activity assessment at the DZHK-examination center.The video can not be skipped.
  Interventions: Other: Video demonstration of physical activity intensity levels
- "No video"-group (No Intervention): No video group: Individuals in this group do not receive the intervention "Video demonstration of physical activity intensity levels". They complete a tablet PC-supported physical activity assessment at the DZHK-examination center without receiving a 3-minute-video explaining and visualizing the different intensity levels of physical activity.

INTERVENTIONS:
Other: Video demonstration of physical activity intensity levels — In the video demonstration, an approximately 50 year old male explains 1) light-intensity, 2) moderate-intensity, and 3) vigorous-intensity physical activity referring to differences in heart rate, breathing frequency and capability to talk normally. Simultaneously, on a treadmill he demonstrates the body signs of the three intensity levels. He gives examples and points out that there are individual differences in the intensity evaluation of comparable activities.
  Arms: "Video"-group

SUMMARY:
This study examines the effect of a video-based intensity level demonstration on self-reported physical activity in individuals aged between 40 and 75 years. Aim of the video demonstration is to achieve a better concordance of physical activity reports with accelerometer-based measurements.

DETAILED DESCRIPTION:
This study examines whether the demonstration of different intensity levels of physical activity by video in the context of a tablet PC (personal computer)-based survey can achieve a higher degree of concordance between self-reported and accelerometer-measured physical activity compared to an assessment without video demonstration. The recruitment of the study participants in the age range between 40 and 75 years takes place in a shopping center in the city Greifswald in Germany.

Informed consent consists of: (i) activity recording over 7 days using an accelerometer, (ii) completion of standardized questionnaires, (iii) participation in a standardized measurement of weight and height as well as waist and hip circumference.

Participants are asked to wear an accelerometer during the day for a period of 7 days. Subsequently, a questionnaire about the frequency, duration and intensity of physical activity in the last 7 days will be answered in the DZHK (Deutsches Zentrum für Herz-Kreislauf-Forschung)- examination center. Prior to the physical activity assessment the study participants are randomly assigned to the study conditions "Video" or "No Video" (ratio 1:1). Optionally, participants may receive feedback on their physical activity measured by accelerometer upon completion of the study.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* cognitive impairment
* inadequate language skills

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Difference between physical activity measured by self-report and by accelerometry | The accelerometer is worn for 7 days and then the IPAQ-SF is retrospectively answered for these 7 days.
  Measures: assessement via tablet PC (International Physical Activity Questionnaire-Short Form, IPAQ-SF) and objective measurement by accelerometry

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Social Medicine and Prevention, University Medicine Greifswald, Greifswald, Germany

REFERENCES:
- [Derived] Voigt L, Ullrich A, Gross S, Guertler D, Jaeschke L, Dorr M, van den Berg N, John U, Ulbricht S. Associations of accelerometer-based sedentary bouts with adiposity markers among German adults - results from a cross-sectional study. BMC Public Health. 2023 Mar 10;23(1):469. doi: 10.1186/s12889-023-15304-8. PMID 36899317